CLINICAL TRIAL: NCT00644020
Title: A Randomized, Double Blind, Placebo Controled, Multicenter Phase ⅡStudy to Evaluate the Safety and Efficacy of Tyroserleutide for Injection in Hepatocellular Carcinoma(HCC) Patients
Brief Title: Phase ⅡStudy of Tyroserleutide for Injection in Hepatocellular Carcinoma(HCC) Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shenzhen Kangzhe Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Xiaoping Chen, Tongji Hospital of Tongji Medical College of HUST
Other Study IDs: TYS-CN-1.1PUMPⅡPartA; TYS-CN-1.1PUMPⅡPartA
Record Dates: First submitted 2008-03-23; First posted 2008-03-26 (Estimated); Last update posted 2008-03-26 (Estimated); Status verified 2007-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — Mitomycin; Fluorouracil

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — collection of blood sample before the operation and ahead of the third and the sixth period.
  collection of the tumor tissue during the operation
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group 1: the Tyroserleutide for injection at the dosage of 3mg/d
  Interventions: Drug: mitomycin, Fluorouracil
- Group 2: the Tyroserleutide for injection at the dosage of 6mg/d
  Interventions: Drug: mitomycin, Fluorouracil
- Group 3: the Tyroserleutide for injection at the dosage of 12mg/d
  Interventions: Drug: mitomycin, Fluorouracil
- Group 4: the placebo group
  Interventions: Drug: mitomycin, Fluorouracil

INTERVENTIONS:
Drug: mitomycin, Fluorouracil — All participants will receive 10mg mitomycin and 1g Fluorouracil through the chemoradiative pump which was transplanted during the operation, and this procedure would be executed a day before each research treatment period.
  Other Names: mitomycin: serial numbers:071006; Fluorouracil: serial numbers:0710071

SUMMARY:
The investigation is a randomized, double-blind, placebo involved and multi-center clinical trial. All subjects are assigned to 4 groups, including 3mg, 6mg, 12mg per day and placebo group. Each group includes 25 subjects, who have hepatic-cellular carcinoma accompanied with branch vein thrombosis. They receive investigational drug 40 days after resection surgery. Each cycle lasts 4 to 6 days with an interval of 29 days in all 6 cycles.

DETAILED DESCRIPTION:
* Patients who have signed the Informed Consent Form and are eligible for the entry criteria will be randomly assigned to either the TYROSERLEUTIDE treatment group or the placebo group. No matter which group the subject is assigned, he/she would receive chemotherapy treatment through the portal vein pump which was transplanted during the carcinoma section surgery 40 days before the randomization.
* Participants will be given either TYROSERLEUTIDE or placebo through intravenous injection with an interval of 29 days, during which the participant will not take any investigational drug or any other anti-tumor treatment as well. On the day just next to the completion of each cycle of research treatment which usually lasts for 3-5 days, the participant will receive medical inspection so as to observe and ensure drug safety.
* Participants will continue to receive investigational drug for 6 cycles until being detected with recurrence or metastasis of tumor or experiencing any serious side effects.
* A CT scan or MRI scan will be performed for each participant to exclude the recurrence or metastasis of tumor and assess the effects of treatment once before the initiation of each new cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age between 18 and 75 years
3. Hepatocellular Carcinoma accompanied with branch vein thrombosis
4. Carcinoma and bolt resection Integrity, cutting edge no tumor cells by microscopic lens in operation
5. CTA or MRI no Carcinoma and bolt after operation

Exclusion Criteria:

1. hypersensitivity to the composition similarity of investigational drug
2. Concomitance other system primary tumor
3. surface area 1.47m2～1.92m2
4. HBV (-) and HCV(-)
5. Patients who have received resectional surgery for HCC
6. HCC complicating main portal vein cork
7. HCC complicating hepatic vein cork
8. Patients who have received systematicness therapy for HCC
9. Patients who have received immunoregulant 4 weeks before randomization
10. Concurrent participation in another clinical trial involving experimental treatment is excluded 4 weeks before randomization
11. uncontrolled infection, hemorrhage, guts leakage postoperative complications
12. postoperative liver function Child-pugh C
13. no evidence of extra-hepatic metastases postoperative
14. no utility sample for gene chip research
15. no physical examination, laboratory and imageology examination that baseline request

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCC complicating branch cork after resection
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-08 (Estimated); Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
DFS(disease free survival) | six month

SECONDARY OUTCOMES:
1.OS （Overall Survival） 2.QOL (quality of life) | six month

CONTACTS AND LOCATIONS:
Overall Officials: Chen X P, Professor, Principal Investigator — Tongji Medical College of Huazhong University of ScienceTechnology
Locations (1):
- A Research Institute of Tumor, Guangzhou, Guangdong, China